CLINICAL TRIAL: NCT06541665
Title: A Multicenter, Phase I, Open-label, Uncontrolled Study of ONO-4059 in Combination With Rituximab, Methotrexate, Procarbazine, and Vincristine (R-MPV) Therapy for Untreated Primary Central Nervous System Lymphoma (PCNSL)
Brief Title: Phase I Study Evaluating Tolerability, Safety, Pharmacokinetics, and Efficacy of Combined ONO-4059 and R-MPV Therapy for PCNSL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4059-13; jRCT2071230124 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Primary Central Nervous System Lymphoma
MeSH Terms: interventions — tirabrutinib; Rituximab; Methotrexate; Procarbazine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tirabrutinib + R-MPV in patients with newly diagnosed, treatment naïve PCNSL (Experimental)
  Interventions: Drug: ONO-4059; Drug: Rituximab; Drug: Methotrexate; Drug: Procarbazine; Drug: Vincristine

INTERVENTIONS:
Drug: ONO-4059 — Specified dose, once daily
  Other Names: Tirabrutinib Hydrochloride
Drug: Rituximab — Specified dose on specified days
Drug: Methotrexate — Specified dose on specified days
Drug: Procarbazine — Specified dose on specified days
Drug: Vincristine — Specified dose on specified days

SUMMARY:
To confirm the tolerability and safety of combined administration of ONO-4059 and R-MPV therapy in untreated PCNSL patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PCNSL
* Patients who have not received treatment for PCNSL in the past
* Patients with ECOG Performance Status 0-2
* Patients expected to survive for 6 months or more

Exclusion Criteria:

* Patients with intraocular PCNSL without brain lesions
* Patients are unable to swallow oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2028-04-28 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Tolerability evaluation | 29 Days
  The number of subjects who experienced adverse events and side effects will be tallied. In the tolerability evaluation part, the number of subjects who experienced Dose Limiting Toxicity(DLT) will be tallied
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) during induction | 2 years
  Adverse events at each visit with the NCI CTCAE v5.0 used as a guide for the grading of severity.

SECONDARY OUTCOMES:
Summary of plasma tirabrutinib concentration at trough and post 2 hours dosing | 30days
Duration of response (DOR) | 2 years
  Duration of response is defined as the time between the date of first response (Complete response (CR), Complete response - unconfirmed (CRu), or partial response (PR) ) and the date of the first progressive disease(PD) according to the IPCG criteria, or date of death due to any cause, whichever occurs first.
Time to response (TTR) | 1 year
  Time to response is defined as the time between the date of first administration of tirabrutinib and the date of first response (CR, CRu, or PR) as determined by IRC according to the IPCG criteria.
Best overall response (BOR) | 1 year
  Best overall response based on independent review committee (IRC) response determination is defined as the best response and is derived programmatically based upon the visit responses determined by IRC from the date of administration of tirabrutinib to the date of PD as determined by IRC or the date of initiation of subsequent anticancer therapy for PCNSL, whichever occurs first.
Complete response rate (CRR) | 4 months
  Complete response rate is defined as the proportion of patients with a best overall response of CR or CRu as determined by an independent review committee according to the IPCG criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (44):
- Japan (44):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Akita University Hospital, Akita, Akita
  - Juntendo University Urayasu Hospital, Urayasu-shi, Chiba
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hospital of the University of Occupational and Environmental Health,Japan, Kitakyushu-shi, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gifu University Hospital (Tokai National Higher Education and Research System), Gifu, Gifu
  - Gunma University Hospital, Maebashi, Gunma
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Hyogo Medical University Hospital, Nishinomiya-shi, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Kanazawa Medical University Hospital, Kahoku-gun, Ishikawa-ken
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - St. Marianna University Hospital, Kawasaki-shi, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Kochi Medical School Hospital, Nankoku-shi, Kochi
  - University of Miyazaki Hospital, Miyazaki, Miyazaki
  - NAGASAKI University Hospital, Nagasaki, Nagasaki
  - Kindai University Nara Hospital, Ikoma-shi, Nara
  - Nara Medical University, Kashihara-shi, Nara
  - Niigata University Medical & Dental Hospital, Niigata, Niigata
  - Oita University Hospital, Yufu-shi, Oita Prefecture
  - Kurashiki Central Hospital, Kurashiki-shi, Okayama-ken
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Saga University Hospital, Saga, Saga-ken
  - Saitama Medical Center, Kawagoe-shi, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Dokkyo Medical University Hospital, Shimotsuga-gun, Tochigi
  - Institute of Science Tokyo Hospital, Bunkyo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - National Hospital Organization Disaster Medical Center, Midorichō, Tokyo
  - The Jikei University Hospital, Minato-ku, Tokyo
  - Toranomon Hospital, Minato-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Toyama University Hospital, Toyama, Toyama
  - Yamaguchi University Hospital, Ube-shi, Yamaguchi
  - University of Yamanashi Hospital, Chuo-shi, Yamanashi

IPD SHARING:
Plan to Share IPD: No